CLINICAL TRIAL: NCT04966598
Title: Using Machine Learning to Predict Acute Kidney Injury in Patients Following Cardiac Surgery
Brief Title: Machine Learning Predict Acute Kidney Injury in Patients Following Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Yunlong Fan (Other)
Responsible Party: Sponsor-Investigator, Yunlong Fan, Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: chinaPLAGH-08983218
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Machine Learning; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is a major complication which may result in adverse impact on short- and long-term mortality. The investigatorshere developed several prediction models based on machine learning technique to allow early identification of patients who at the high risk of unfavorable kidney outcomes.

The retrospective study comprised 2108 consecutive patients who underwent cardiac surgery from January 2017 to December 2020.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years who underwent cardiac surgery

Exclusion Criteria:

* data miss greater than 10%

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: age over 18 years who underwent cardiac surgery
Sampling Method: Probability Sample
Enrollment: 2108 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | 7 days
  postoperative AKI was defined according to KDIGO criteria during the first 7 days after operation. Postoperative AKI was defined as either at an increase of at least 50% within 7 days or 0.3 mg/dL elevation within 48 h compared with the reference serum creatinine level.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shao J, Liu F, Ji S, Song C, Ma Y, Shen M, Sun Y, Zhu S, Guo Y, Liu B, Wu Y, Qin H, Lai S, Fan Y. Development, External Validation, and Visualization of Machine Learning Models for Predicting Occurrence of Acute Kidney Injury after Cardiac Surgery. Rev Cardiovasc Med. 2023 Aug 9;24(8):229. doi: 10.31083/j.rcm2408229. eCollection 2023 Aug. PMID 39076716